CLINICAL TRIAL: NCT01905306
Title: Clinical Evaluation of Immediate Loading Full Arch Rehabilitation Made With Methodology for Computer Guided Implant Planning With Software Polyvalent vs Free Hand Implants Placement
Brief Title: Randomized Controlled Trial of Full-Arch Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Prof. Marco Ferrari, Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCTGIS1; RCTGIS1s (Other: University of Siena)
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Bone-to-implant Contact; Success Rate; Survival Rate
Keywords: dental implants; immediate loading; full-arch; computer guided implant surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- computer guided implant planning (Experimental): radiographic and clinical evaluation of full-arch dental implant rehabilitation
  Interventions: Procedure: computer guided implant planning
- free hand implants placement (Experimental): radiographic and clinical evaluation of full-arch dental implant rehabilitation
  Interventions: Procedure: free hand implants placement

INTERVENTIONS:
Procedure: computer guided implant planning
  Arms: computer guided implant planning
Procedure: free hand implants placement
  Arms: free hand implants placement

SUMMARY:
This clinical study has the objective to compare the radiographic evaluations after 3 years of follow-up of immediate loaded implant-prosthetic rehabilitation, carried out randomly using the methodology for computer guided implant planning with software polyvalent or free hand implants placement.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous patients with an adequate area: at least two teeth in the posterior area
* Age over 18 years
* Adequate width of the bone crest without the need for bone regeneration
* Consensus to participate in a oral hygiene maintenance program
* Consensus to participate in a long-term study
* Availability to provide their free and informed consensus.

Exclusion Criteria:

* Systemic diseases that preclude participation in the study
* History of radiation therapy
* Bone lesions
* Cigarette smoking (more than 10 cigarettes per day)
* Inadequate oral hygiene
* Untreated periodontitis affecting residual teeth

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
bone-to-implant contact | 3 years
  2D radiographic assessment of the implant surface in contact with bone expressed in percentage

SECONDARY OUTCOMES:
implant survival rate | 3 years
  1. the absence of clinically detectable implant mobility
  2. a lack of persistent or irreversible signs and symptoms such as pain or any subjective sensation
  3. the absence of recurrent peri-implant infection
  4. the absence of concrete evidence of continuous periimplant radiolucency

OTHER OUTCOMES:
implant success rate | 3 years
  1. No pain or tenderness upon function
  2. 0 mobility
  3. 2 mm radiographic bone loss from initial surgery
  4. No exudates history

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ferrari, Prof, Principal Investigator — University of Florence and Siena, Siena, Italy
Locations (1):
- Department of Dental Materials and Fixed Prosthodontics of Siena, Tuscan School of Dental Medicine, University of Florence and Siena, Siena, Siena, Italy

REFERENCES:
- [Background] Drago C, del Castillo R, Peterson T. Immediate occlusal loading in edentulous jaws, CT-guided surgery and fixed provisional prosthesis: a maxillary arch clinical report. J Prosthodont. 2011 Apr;20(3):209-17. doi: 10.1111/j.1532-849X.2010.00661.x. Epub 2010 Nov 11. PMID 21070431
- [Background] Case study: computer-guided implant successful in high-risk patient. J Calif Dent Assoc. 2012 Oct;40(10):784. No abstract available. PMID 23316558
- [Background] Margonar R, Queiroz TP, Luvizuto ER, Santos PL, Wady AF, Paleari AG. Anterior tooth rehabilitation with frozen homogenous bone graft and immediately loaded titanium implant using computer-guided surgery. J Craniofac Surg. 2012 Sep;23(5):e470-2. doi: 10.1097/SCS.0b013e3182587516. PMID 22976712
- [Background] Nickenig HJ, Eitner S, Rothamel D, Wichmann M, Zoller JE. Possibilities and limitations of implant placement by virtual planning data and surgical guide templates. Int J Comput Dent. 2012;15(1):9-21. English, German. PMID 22930944
- [Background] Shibly O, Kutkut A, Albandar JM. One-year re-entry results of guided bone regeneration around immediately placed implants with immediate or conventional loading: a case series. J Int Acad Periodontol. 2012 Jul;14(3):62-8. PMID 22908535
- [Background] Schnitman PA, Lee SJ, Campard GJ, Dona M. Guided flapless surgery with immediate loading for the high narrow ridge without grafting. J Oral Implantol. 2012 Jun;38(3):279-88. doi: 10.1563/AAID-JOI-D-11-00215. PMID 22783940